CLINICAL TRIAL: NCT07309640
Title: The Effects of Magnesium (Mg) Supplement and Alternate Maxillary Expansion and Constriction (Alt-RAMEC) in Patient With Transverse Maxillary Deficiency (TMD): A Randomized Clinical Trial.
Brief Title: The Effects of Magnesium (Mg) Supplement and Alternate Maxillary Expansion and Constriction (Alt-RAMEC) in Patient With Transverse Maxillary Deficiency (TMD)
Acronym: Mg + Alt-RAMEC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, IBRAHEEM RAHMA HAZIM IBRAHEEM, principle invistegator, Universiti Sains Malaysia
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: USM/JEPeM/KK/24070610
Record Dates: First submitted 2025-11-30; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Magnesium During Orthodontic Expansion; Orthodontic Patients Indicated for Maxillary Expansion
Keywords: Expansion; Magnesium; Orthodontic
MeSH Terms: interventions — magnesium citrate; Magnesium

STUDY DESIGN:
Intervention Model Description: Model Description for the Interventional Study Model (Parallel Assignment):
  This randomized clinical trial utilizes a parallel assignment design in which adult patients with transverse maxillary deficiency are randomly allocated into two groups. One group receives the Alternate Maxillary Expansion and Constriction (Alt-RAMEC) protocol using the Micro-implant Assisted Rapid Palatal Expansion (MARPE) appliance alone, while the second group receives the same protocol combined with oral magnesium supplementation.
  Both groups undergo the interventions simultaneously but independently, allowing comparison of the outcomes related to dental, skeletal, muscular, and patient-reported factors. The parallel design facilitates the evaluation of the added effect of magnesium supplementation on the efficacy and patient experience during the orthodontic expansion treatment.
  This design supports unbiased comparison between intervention effects in two distinct groups treated concurrently.
Masking Description: Masking Description:
  There are no additional parties masked in this clinical trial. The study is conducted as an open-label trial with no blinding of participants, investigators, or outcome assessors. All parties are aware of the treatment assignments throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control group (Other): Normal expansion activities
  Interventions: Dietary Supplement: magnesium citrate; Dietary Supplement: Magnesium

INTERVENTIONS:
Dietary Supplement: magnesium citrate — using in orthodontic patients
Dietary Supplement: Magnesium — Mg supplement provoke more sutural separation and bone integrity (density and thickness) in Alt-Ramec protocol compared to the normal expansion protocol?

SUMMARY:
This randomized clinical trial evaluates the effect of combining magnesium supplementation with an orthodontic technique called Alternate Maxillary Expansion and Constriction (Alt-RAMEC) using a Micro-implant Assisted Rapid Palatal Expansion (MARPE) appliance to treat adults (18-30 years) with transverse maxillary deficiency (TMD). TMD is a condition where the upper jaw is narrower than normal, which can affect bite and facial development.

The study involves two groups: one receiving the Alt-RAMEC protocol with MARPE alone, and the other receiving the same protocol alongside oral magnesium supplements. The effectiveness of these treatments will be compared by assessing changes in dental and skeletal structures through imaging techniques and evaluating muscle function. Participants will also report their pain and discomfort levels during the treatment.

This research aims to understand whether magnesium supplementation can enhance the effects of Alt-RAMEC treatment, improve patient outcomes, and reduce discomfort associated with orthodontic procedures.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the effectiveness of magnesium supplementation combined with the Alternate Maxillary Expansion and Constriction (Alt-RAMEC) protocol using Micro-implant Assisted Rapid Palatal Expansion (MARPE) in adult patients with transverse maxillary deficiency (TMD). The study compares two treatment groups: one receiving the Alt-RAMEC protocol with MARPE alone, and the other receiving Alt-RAMEC with MARPE alongside oral magnesium supplementation.

The Alt-RAMEC protocol involves controlled cycles of maxillary expansion and constriction to facilitate the correction of maxillary transverse discrepancies. Patients are treated with specific activation and deactivation regimens involving the MARPE appliance over several weeks. This study assesses changes in dental, alveolar, skeletal, and muscular structures by using advanced imaging such as 3D Cone Beam Computed Tomography (CBCT) and surface electromyography (sEMG). Additionally, patient-reported pain and discomfort levels will be evaluated during the orthodontic treatment.

This trial focuses on objectively measuring morphological and functional changes to determine whether magnesium intake enhances the effects of the Alt-RAMEC treatment and improves patient comfort and treatment outcomes. The findings may provide valuable evidence for optimizing management protocols for transverse maxillary deficiency in young adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. All participants were young adults, from the 18- 25 age group (males or females).
  2. There is a maxillary skeletal deficiency in every patient. (Anteroposterior deficiency, transverse bilateral/unilateral deficiency)
  3. All teeth erupted without any abnormalities in term of shape and size.
  4. Good oral hygiene and non-smoking habits.

Exclusion Criteria:

1. History of previous orthodontic treatment or maxillary expansion
2. Patients with severe progressive periodontal disease
3. Patients with severe craniomaxillofacial deformities such as cleft lip and palate
4. Mid palatal fusion without successful expansion
5. First molar absent or impacted in the patient.
6. Patients who have bone loss, gingival recession, or persistent gingival inflammation.
7. Individuals with a high gag reflex.
8. History of a life-threatening medical condition, such as diabetes mellitus, or a chronic disease such as organ transplant rejection or cancer in patients receiving chemotherapy or radiation therapy and high risk of infections.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-12 (Estimated); Study Completion 2026-09-12 (Estimated)

PRIMARY OUTCOMES:
The Primary Outcome Measure title for this clinical study is: Change in Transverse Maxillary Dimensions and Muscular Activity Following Alt-RAMEC Protocol with or without Magnesium Supplementation | The Time Frame for the primary outcome measure in this clinical trial is: Pre-treatment (T0) to Post-treatment (T1), including the active expansion period after 12 weeks of alternate expansion and constriction
  Primary Outcome Description:
  The primary outcome of this study is to assess the changes in transverse maxillary dimensions and muscular activity in adult patients with transverse maxillary deficiency following treatment with the Alternate Maxillary Expansion and Constriction (Alt-RAMEC) protocol using Micro-implant Assisted Rapid Palatal Expansion (MARPE) with or without magnesium supplementation.
  This includes quantitative measurements of skeletal and dentoalveolar changes using 3D Cone Beam Computed Tomography (CBCT) imaging, evaluation of muscular changes via surface electromyography (sEMG) during dental clench and chewing, and assessment of patient-reported pain and discomfort using a visual analog scale. The study compares these parameters pre-treatment (T0) and post-treatment (T1) to determine the efficacy and effects of the interventions on maxillary expansion and muscular adaptations.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine IBSU University, Baghdad , Iraq, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared outside the research team due to concerns related to protecting patient confidentiality and privacy. The data contains sensitive health information, and sharing it could pose risks despite de-identification efforts. Additionally, data sharing is subject to ethical approvals and agreements that limit dissemination to safeguard participants' rights. This restriction ensures compliance with institutional, ethical, and legal standards governing participant data security.